CLINICAL TRIAL: NCT07381231
Title: A Prospective Phase II Study of Immunotherapy With Adaptive Pulse Radiotherapy in Solid Tumors
Brief Title: Immunotherapy With Adaptive Pulse Radiotherapy in Solid Tumors
Acronym: I-APT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Nalee Kim, Assistant professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2025-08-014; 2025-08-014 (Other: Samsung medical center)
Record Dates: First submitted 2025-12-01; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Immunotherapy; Radiation therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulse RT (Experimental)
  Interventions: Radiation: Pulse radiation therapy

INTERVENTIONS:
Radiation: Pulse radiation therapy — Adaptive Pulse Radiotherapy (Pulse RT) is a personalized radiotherapy strategy designed to enhance anti-tumor immunity when combined with immune checkpoint inhibitors (ICIs). Patients receive 2-3 fractions of 8-10 Gy at 3-4-week intervals, with adaptive modification of target volumes according to tumor response. This approach aims to induce repeated immunogenic cell death and expand tumor-specific T-cell repertoires, thereby amplifying the efficacy of concurrent immunotherapy while maintaining safety within standard dose constraints. Both photon and proton modalities may be used, depending on lesion location and clinical judgment.

SUMMARY:
The goal of this clinical trial is to find out whether Adaptive Pulse Radiotherapy (Pulse RT) combined with immune checkpoint inhibitors (ICIs) helps treat advanced solid tumors.

It will also check how safe this combined treatment is and how it affects the immune system and quality of life.

The main questions the study will try to answer are:

Does adding Pulse RT to ICIs improve tumor response and survival? What side effects occur when participants receive Pulse RT with ICIs? How does the treatment change immune-related blood and tissue markers? Does the treatment affect participants' quality of life?

Researchers will compare this new approach to usual ICI treatment to see whether Pulse RT makes a difference.

Participants will:

Continue to receive their standard ICI treatment. Receive 2-3 sessions of high-dose Pulse RT (8-10 Gy each) given about every 3 weeks.

Have the treatment volume adjusted based on how their tumors respond. Visit the clinic regularly for check-ups, imaging, blood tests, and quality-of-life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Histologically confirmed solid tumor (radiologic diagnosis allowed for hepatocellular carcinoma)
* Currently receiving or planned to receive immune checkpoint inhibitor (ICI) therapy
* Presence of at least one lesion suitable for radiotherapy and measurable disease per RECIST version 1.1
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Presence of brain metastasis or leptomeningeal metastasis
* Prior radiotherapy to the intended treatment site
* Significant comorbid conditions that may interfere with study participation or treatment (e.g., uncontrolled infection, heart failure, arrhythmia, psychiatric disorder)
* Inability or unwillingness to comply with study procedures
* Considered inappropriate for study participation by the principal investigator or treating physician

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival at 6 Months | 6 months after first radiation therapy
  Progression-free survival (PFS) is defined as the time from the start of Adaptive Pulse Radiotherapy (first radiation treatment) to the date of disease progression according to RECIST version 1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 3, 6, 12, 24, and 36 months after initiation of Adaptive Pulse Radiotherapy
  Progression-free survival (PFS) will be assessed using Kaplan-Meier analysis.
Local Recurrence-Free Survival (LRFS) | 3, 6, 12, 24, and 36 months after initiation of Adaptive Pulse Radiotherapy
  Local recurrence-free survival (LRFS) is defined as the time from initiation of Adaptive Pulse Radiotherapy to local tumor recurrence within the irradiated field or death from any cause, whichever occurs first.
Overall Survival (OS) | 3, 6, 12, 24, and 36 months after initiation of Adaptive Pulse Radiotherapy
  Overall survival (OS) is defined as the time from initiation of Adaptive Pulse Radiotherapy to death from any cause.
Objective Response Rate (ORR) | 3, 6, 12, 24, and 36 months after initiation of Adaptive Pulse Radiotherapy
  Objective response rate is defined as the proportion of participants achieving complete or partial response according to RECIST version 1.1 criteria.
Immune Response Profiling and Biomarker Analysis | Baseline, during treatment, 1 month after last radiation therapy
  Changes in circulating immune biomarkers, including cytokine levels (e.g., IL-6, IL-8, IL-10, TNF-β, IFN-γ) and immune cell subsets (e.g., CD3, CD4, CD8, NK cells, regulatory T cells), will be assessed in peripheral blood samples collected at specified time points.
Change in Patient-Reported Quality of Life | Baseline, During treatment, 3, 6, 12, 24, and 36 months after initiation of Adaptive Pulse Radiotherapy
  Patient-reported outcomes will be evaluated using the PRO-CTCAE core set at baseline and during follow-up. Changes over time will be analyzed using linear mixed models to assess treatment-related symptom burden and overall quality of life trends.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided